CLINICAL TRIAL: NCT02132442
Title: Hepatic Dysfunction, Vitamin D Status, and Glycemic Control in Diabetes
Acronym: VDLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Benjamin U. Nwosu, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC Docket # H00002866
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes; Nonalcoholic Fatty Liver Disease; Vitamin D Deficiency
Keywords: Children; Adolescents; Adults; Type 2 diabetes; Nonalcoholic fatty liver disease; Vitamin D deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D supplementation (Experimental): Ergocalciferol 50,000 IU per week for 6 weeks, then bi-weekly for 6 mo
  Interventions: Dietary Supplement: Ergocalciferol, placebo
- Placebo (Placebo Comparator): Placebo capsules, on capsule per week for 6 weeks, then bi-weekly for 6 mo.
  Interventions: Dietary Supplement: Ergocalciferol, placebo

INTERVENTIONS:
Dietary Supplement: Ergocalciferol, placebo — Ergocalciferol 50000 IU capsules Microcrystalline cellulose
  Other Names: Vitamin D; Placebo

SUMMARY:
This study is designed to study the effect of vitamin D intake on the severity of fatty liver and poor glucose control in patients with type 2 diabetes and fatty liver disease.

DETAILED DESCRIPTION:
The prevalence of significantly poor glycemic control marked by a hemoglobin A1c (HbA1c) level of ≥ 9.5% in youth with type 2 diabetes (T2D) is 27% 1 and 24.2% in young adults2. Strategies to improve glycemic control in patients with T2D include lifestyle modification, optimization of therapeutic regimens, and correction of comorbid states that impair glycemic control. However, the role of comorbid states on glycemic control in T2D has not been adequately studied. For example, 70% of patients with T2D have nonalcoholic fatty liver disease (NAFLD)3, a potentially serious form of chronic liver disease 4 in which the triad of the development of lipotoxicity-induced mitochondrial dysfunction, activation of inflammatory pathways, and cytokine generation lead to progressive liver damage5. NAFLD is the leading cause of elevated liver enzymes in the US6, and is diagnosed by either liver biopsy or the detection of a hepatic triglyceride content (HTGC) of >5.6% by proton magnetic resonance spectroscopy (1H MRS)2. Despite the high prevalence of NAFLD in T2D, its potential impact on glycemic control through the impairment of hepatic metabolic processes is unclear. This is important because a crucial step in vitamin D metabolism, the hydroxylation of vitamin D at the 25 position, occurs in the liver. The consequence of NAFLD on this critical step in vitamin D metabolism in patients with T2D, and the impact of the resultant 25-hydroxyvitamin D [25(OH)D] deficiency on glycemic control are not well understood. The rationale for this study is that a clear understanding of the role of vitamin D on the pathogenesis of NAFLD is crucial because vitamin D is a prohormone with potent anti-inflammatory properties that inhibit pro-inflammatory cytokines such as tumor necrosis factor- α (TNF-α), interleukin-6, and the activity of macrophages 2 while upregulating the production of anti-inflammatory cytokine, interleukin-10 2which could potentially reverse the effects of insulin resistance (IR) and oxidative stress, the two key components of the 'double hit model' of the pathogenesis of NAFLD. The 'first hit' involves IR-induced hepatocyte lipid accumulation which increases hepatic vulnerability to the components of the 'second hit': oxidative stress and proinflammatory cytokines, leading to mitochondrial dysfunction, inflammation and fibrosis.

The investigators7 previously showed that mild hepatic dysfunction in patients with T2D was associated with a high prevalence (47.5%) of vitamin D deficiency as defined by 25(OH)D level of < 20 ng/mL, as well as poor glycemic control. The investigators further reported a significant inverse relationship between HbA1c and 25(OH)D, and also between 25(OH)D and alanine transaminase. These data suggest that mild hepatic dysfunction could impair vitamin D metabolism and negatively impact glycemic control in patients with T2D. The investigators have also accumulated data 8 to show that 25(OH)D supplementation was associated with a significant reduction in HbA1c in T2D without a significant change in insulin or metformin dose. Histologically, a recent animal study reported significant hepatic steatosis in vitamin D-deficient mice compared to vitamin D-sufficient mice 2.

ELIGIBILITY:
Inclusion Criteria:

1. Children: 10 - 17 years
2. Adults: 18 - 50 years
3. Type 2 diabetes > 6 mo duration
4. 25-hydroxyvitamin D [25(OH)D] level of <20 ng/mL
5. Hepatic triglyceride content (HTGC) value of >5.6%
6. HbA1c of > 8%;
7. Ability to take medication by mouth.

Exclusion Criteria:

1. Pregnant or lactating women
2. Mental deficiency (IQ <70)
3. Chronic liver disease
4. Disorders of vitamin D metabolism, kidney, or parathyroid disease;
5. Calcium and/or vitamin D supplementation
6. Mauriac syndrome
7. Malabsorption of fat soluble vitamins
8. Drug toxicity and alcoholism

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in hepatic triglyceride content (HTGC) | 6 months
  Change in hepatic triglyceride content (HTGC) as measured by proton magnetic resonance spectroscopy (1H MRS)

SECONDARY OUTCOMES:
Hemoglobin A1c | 6 months
  Change in glycemic control as measured by HbA1c.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States